CLINICAL TRIAL: NCT04882267
Title: General Health, Attitudes, and Activity in Self-directed Exercise in Patients With Cystic Fibrosis (GAINS-CF)
Acronym: GAINS-CF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Lindsay Somerville, MD, Associate Director of Adult CF Medicine, University of Virginia
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: HSR200451-GAINS-CF
Record Dates: First submitted 2021-05-07; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Cystic Fibrosis
Keywords: exercise; cystic fibrosis; CF; mental health
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity; Psychological Well-Being | interventions — Technology

STUDY DESIGN:
Intervention Model Description: Subjects will serve as own controls to establish a baseline of physical activity (first arm). After the baseline period, subjects will partake in the 4-week intervention in which they receive access to home exercise apps and receive motivational interviewing phone calls (second arm). After the intervention period, subjects will continue to have access to apps, but no longer receive phone calls. Activity and surveys will be measured at the end of 4 weeks (third arm).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Determination of attitudes and perceived barriers to exercise (No Intervention): Adults with CF will take part in a quantitative modified Exercise Benefits/Barriers Scale (EB/BS) survey to identify universal and unique benefits and barriers to regular exercise activity. Subjects will be surveyed on potential ways to engage in exercise, including perceptions and prior use of smart device exercise technology. Qualitative input will be incorporated to better understand potential solutions to barriers, and develop more personalized plans for exercise engagement.
- Determination of baseline exercise activity (Baseline Period) (No Intervention): Adults with CF who identify as 'willing to use technology' and own compatible smart phones/tablets will undergo the Short General Health Questionnaires (GHQ 12) to establish baseline levels of general and mental health. Subjects will be fitted with wrist actigraphy and monitored for four weeks to establish baseline levels of exercise activity at home. Anticipated outcomes: Access to actigraphy will encourage personal accountability, and physical activity will increase during the first two weeks before reaching a plateau.
- Engagement in home self-directed exercise incorporating Team and Technology (Intervention Period) (Experimental): Subjects will take part in a live demonstration of three subscription-based AI-learning home exercise apps, and one self-directed exercise website designed by a CF patient partner. Subjects will be surveyed on willingness to use technology, and provide feedback on exercise options. They will be given free full access to the apps and website ("Technology"), and receive a phone call once a week from their CF specialty team offering encouragement and positive reinforcement ("Team"). App and website usage, actigraphy, EB/BS and GHQ 12 scores will be measured at the end of four weeks. Anticipated outcomes: Activity will increase significantly during the Team and Technology intervention period, barriers on the EB/BS score will decrease, and GHQ 12 scores will increase.
  Interventions: Behavioral: Team and Technology
- Determination of sustainability (Sustainability Period) (Active Comparator): Phone calls will cease, but subjects will maintain access to apps, websites, and actigraphy. After four weeks, EB/BS and GHQ 12 scores, physical activity, app and website use will be reassessed. Anticipated outcomes: Activity will decrease during the sustainability period, but will remain significantly greater than the pre-intervention period. Overall GHQ 12 and EB/BS scores will improve.
  Interventions: Behavioral: Team and Technology

INTERVENTIONS:
Behavioral: Team and Technology — Subjects will receive access and instruction on multiple home exercise apps. They will receive phone calls once a week from care team members for motivational interviewing to encourage exercise.
  Arms: Determination of sustainability (Sustainability Period); Engagement in home self-directed exercise incorporating Team and Technology (Intervention Period)

SUMMARY:
Exercise helps people with CF lead long, fulfilling lives. Regular exercise reduces depression and fatigue, and may play a role in preventing exacerbation. However, little is known about exercise habits in adults with CF, or the barriers to exercise that they face.

During the COVID-19 pandemic, lockdowns and social distancing saw gym memberships plummet; while sale of personal exercise technology, smart-watches, and interactive home equipment exploded. As this technology becomes more cost-effective and accessible, can it be leveraged to improve CF care? This study will examine barriers to exercise in CF and the role of smart devices in exercise. Adults with CF will participate in the Exercise Behaviors/Barriers Survey, followed by a qualitative discussion on attitudes toward exercise technology, and how CF impacts exercise. We anticipate that many perceived barriers will be universal (e.g. time), while others will be unique to CF.

Participants will be fitted with wrist actigraphy (FitBit Inspire 2) to measure baseline exercise. They will receive access to three smartphone apps designed for home exercise, as well as an exercise website designed for the CF community (www.activate65.org), and receive weekly phone calls from the CF care team offering motivational interviewing. Actigraphy, heart and respiratory rate, and app usage will be analyzed. After four weeks, participants will no longer receive calls. Actigraphy will be monitored four additional weeks to determine if exercise is sustained. We anticipate that exercise will increase during the intervention period, and that some activity will be sustained in the follow up period.

The findings of this study will pave the way for a larger trial using this "Team and Technology" approach to investigate clinical outcomes. This study highlights the critical and timely need to investigate the barriers to exercise in CF, and effective solutions to develop sustainable exercise habits using widely-available technology from home.

DETAILED DESCRIPTION:
Adults with CF aged 18 and above, who have access to either Google Play (Google LLC) or Apple (Apple Inc.) smart device, and are patients of the University of Virginia Adult CF clinic will be enrolled in this study. Subjects will be invited by the PI during routine pre-visit planning for quarterly appointments. Subjects who are unable to provide consent, pregnant or trying to become pregnant, or have a known physical condition that precludes exercise will be excluded. Enrolled subjects will serve as their own controls, and there will be an additional four healthy non-CF controls. We will recruit subjects from each lung function subgroup FEV1 < 40%, FEV1 40-79%, and FEV1 >80%.

Enrolled subjects will be screened using the Physical Activity Readiness Questionnaire (PAR-Q) prior to exercise. Respondents who are not eligible for exercise based on PAR-Q results will be excluded. Subjects will participate in the Exercise Benefits/Barriers Scale (EB/BS) to identify perceived benefits and barriers to exercise via online secured Qualtrics Research Suite link. They will participate in a one-on-one conversation with the PI answering open-ended questions about how their life experience with CF may impact exercise behavior, as well as their attitudes toward use of personal technology in exercise. Input will be qualitatively analyzed for themes that may aid in developing more personalized plans for exercise engagement.

Subjects will complete the Short General Health Questionnaire (GHQ 12) to establish self-reported baseline levels of general physical and mental health. They will be fitted with a wrist actigrapher (FitBit Inspire 2; Google, LLC). They will receive training on FitBit usage and how to safely export data via HIPAA-secured electronic communication. For four weeks, physical activity will be logged, including steps per day, time spent in aerobic activity, respiratory rate, and heart rate. This will establish baseline levels of activity.

Subjects will then begin the "Team & Technology" exercise intervention. Team: Participants will receive weekly phone calls from members of the CF care team encouraging exercise and offering motivational interviewing personalized from earlier interviews. Technology: Participants will take part in a live demonstration of three subscription-based exercise apps compatible with Apple and Google Play personal devices, and will receive unlimited access to all apps. They will also receive access to a mobile-friendly exercise community website designed by UVA patient partner for adults with CF (www.activate65.org, Elize Hewitt, 2021). The apps were selected based of their ability to provide a variety of workouts from home using only body weight, without specialized equipment. Apps included in this study are BodBot (BodBot, LLC), an AI-learning exercise app that customizes exercise plans to the user and incorporates body weight and aerobic exercise; SHRED (Shred Labs, LLC), an AI-learning exercise app that incorporates both muscle-building and aerobic exercise; Seven (Perigee AB), and J&J Official 7 Minute Workouts (Johnson & Johnson Health and Wellness Solutions, Inc) two apps that generate high-intensity interval training (HIIT) workouts in 7-minute intervals based on self-selected skill level. Subjects will be encouraged to exercise using any method they wish, including using any combination of the technology options, or their own methods. Multiple apps with different methods and styles have been selected so that any one specific app does not become the intervention per se, but rather provides exercise options. Physical activity will be logged, along with app and website usage. After four weeks, EB/BS and GHQ 12 surveys will be repeated.

After the intervention period, motivational phone calls will end. Subjects will still have unlimited access to the technology, and will continue to wear actigraphers. Technology usage and physical activity will be logged at the end of an additional four weeks to assess for sustainability of exercise habits. Finally, EB/BS and GHQ 12 surveys will be repeated during a debrief phase.

This pilot study will identify perceived benefits and barriers to exercise, based on the unique lived experiences of adults with CF. We will determine whether attitudes toward exercise correlate with elements of emotional and physical wellbeing, and we will assess whether perceived benefits and barriers toward exercise can be positively shaped by motivational interviewing and encouragement from the individual's care team. We will further determine whether the use of widely available personal smart devices can be leveraged to form sustainable exercise habits in adults with CF.

Exercise is a critical component to physical and mental health, and is of particular importance as we inch closer to a cure for CF. We believe that the qualitative input on attitudes toward exercise behavior will be a valuable aspect to creating sustainable exercise plans that address the specific challenged faced by people with CF. We hypothesize that having access to wrist actigraphy alone will increase physical activity by creating immediate positive feedback and personal accountability. We further anticipate that having access to a variety of home workout options, along with personal support and motivational interviewing from the CF care team, will increase overall exercise habits and positively impact attitudes toward exercise. We hypothesize that physical activity will decrease in the sustainability period, but overall activity and attitudes toward perceived barriers will improve compared to baseline.

If exercise sustainability is observed as we anticipate, we plan to embark on a large, randomized controlled using pilot data to inform power analysis. This trial will investigate the role of sustained home exercise in CF on lung function, exacerbation rates, mental health, BMI, lean muscle composition, and other important clinical outcomes. These questions are of particular interest in the era of highly-efficacious CFTR modulator therapies that are extending length and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Must have access to either Google Play (Google LLC) or Apple (Apple Inc.) smart device
* Patients of the University of Virginia Adult CF clinic

Exclusion Criteria:

* Unable to exercise based on PAR-Q survey
* Known physical condition that precludes exercise
* Pregnant, or trying to become pregnant
* Unable to provide informed consent
* Prisoners
* Does not own and feel comfortable using a smart device
* Unwilling to use smart devices for research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-05-31 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Activity levels | ten weeks
  Activity measured in steps per day
Activity levels | ten weeks
  Activity measured by heart rate above target in minutes per day
Perceived barriers and benefits of exercise | ten weeks
  Perceived barriers and benefits of exercise as measured by serial EB/BS surveys
General and Mental Health | ten weeks
  General and mental health scores as measured by the GHQ 12

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Somerville, MD, Principal Investigator — University of Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nixon PA, Orenstein DM, Kelsey SF, Doershuk CF. The prognostic value of exercise testing in patients with cystic fibrosis. N Engl J Med. 1992 Dec 17;327(25):1785-8. doi: 10.1056/NEJM199212173272504. PMID 1435933
- [Background] Hulzebos EH, Bomhof-Roordink H, van de Weert-van Leeuwen PB, Twisk JW, Arets HG, van der Ent CK, Takken T. Prediction of mortality in adolescents with cystic fibrosis. Med Sci Sports Exerc. 2014 Nov;46(11):2047-52. doi: 10.1249/MSS.0000000000000344. PMID 24848493
- [Background] Sharma R, Florea VG, Bolger AP, Doehner W, Florea ND, Coats AJ, Hodson ME, Anker SD, Henein MY. Wasting as an independent predictor of mortality in patients with cystic fibrosis. Thorax. 2001 Oct;56(10):746-50. doi: 10.1136/thorax.56.10.746. PMID 11562511
- [Background] Orava C, Fitzgerald J, Figliomeni S, Lam D, Naccarato A, Szego E, Yoshida K, Fox P, Sykes J, Wu K. Relationship between Physical Activity and Fatigue in Adults with Cystic Fibrosis. Physiother Can. 2018;70(1):42-48. doi: 10.3138/ptc.2016-75. PMID 29434417
- [Background] Carek PJ, Laibstain SE, Carek SM. Exercise for the treatment of depression and anxiety. Int J Psychiatry Med. 2011;41(1):15-28. doi: 10.2190/PM.41.1.c. PMID 21495519
- [Background] Shelley J, Boddy LM, Knowles ZR, Stewart CE, Dawson EA. Physical activity and associations with clinical outcome measures in adults with cystic fibrosis; a systematic review. J Cyst Fibros. 2019 Sep;18(5):590-601. doi: 10.1016/j.jcf.2019.03.003. Epub 2019 Mar 27. PMID 30926321
- [Background] Jantzen A, Opoku-Pare M, Bieli C, Ruf K, Hebestreit H, Moeller A. Perspective on cystic fibrosis and physical activity: Is there a difference compared to healthy individuals? Pediatr Pulmonol. 2016 Oct;51(10):1020-1030. doi: 10.1002/ppul.23532. Epub 2016 Jul 26. PMID 27459056
- [Background] Thomson RL, Buckley JD, Brinkworth GD. Perceived exercise barriers are reduced and benefits are improved with lifestyle modification in overweight and obese women with polycystic ovary syndrome: a randomised controlled trial. BMC Womens Health. 2016 Mar 9;16:14. doi: 10.1186/s12905-016-0292-8. PMID 26960762
- [Background] Anjara SG, Bonetto C, Van Bortel T, Brayne C. Using the GHQ-12 to screen for mental health problems among primary care patients: psychometrics and practical considerations. Int J Ment Health Syst. 2020 Aug 10;14:62. doi: 10.1186/s13033-020-00397-0. eCollection 2020. PMID 32793301
- [Background] Rovedder PM, Flores J, Ziegler B, Casarotto F, Jaques P, Barreto SS, Dalcin Pde T. Exercise programme in patients with cystic fibrosis: a randomized controlled trial. Respir Med. 2014 Aug;108(8):1134-40. doi: 10.1016/j.rmed.2014.04.022. Epub 2014 Jun 26. PMID 25002195